CLINICAL TRIAL: NCT00033345
Title: Multiple Daily Dose Phase I Safety And Pharmacokinetic Clinical Study Of Indole-3-Carbinol
Brief Title: Indole-3-Carbinol in Preventing Breast Cancer in Nonsmoking Women Who Are at High Risk For Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KUMC-8508-01; CDR0000069276 (Registry Identifier: PDQ (Physician Data Query)); NCI-P02-0217
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — indole-3-carbinol

ARMS (1):
- High-Risk Breast Cancer (Experimental): All subjects first went through a 4-week placebo run-in period. Next, subjects took Indole-3-carbinol 400mg daily for 4 weeks followed by a 4-week period of Indole-3-carbinol 800mg daily.
  Interventions: Drug: Indole-3-carbinol; Other: Placebo

INTERVENTIONS:
Drug: Indole-3-carbinol — 400 mg pill taken daily
  Other Names: I3C
Drug: Indole-3-carbinol — 800 mg pill taken daily
  Other Names: I3C
Other: Placebo — Placebo pill taken daily during run-in period

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Indole-3-carbinol may be effective in preventing breast cancer.

PURPOSE: Phase I trial to study the effectiveness of indole-3-carbinol in preventing breast cancer in nonsmoking women who are at high risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of indole-3-carbinol for the prevention of breast cancer in non-smoking women at high risk for breast cancer.
* Determine the pharmacokinetics of this drug in these participants.
* Determine the effect of this drug on metabolites of estrogen in urine of these participants.
* Determine other additional effects of this drug on selected indicators of drug metabolism and reproductive and hormonal function in these participants.
* Assess any possible antineoplastic activity of this drug in these participants.
* Determine the quality of life of participants receiving this drug.

OUTLINE: This is a single-blind study.

Participants ingest study compound twice daily on weeks 1-12 or 1-16. Study compound is dispensed on weeks 1, 5, and 9. At times, study compound is oral placebo, and at other times, oral indole-3-carbinol.

Quality of life is assessed at baseline and then every 4 weeks during study therapy.

PROJECTED ACCRUAL: A total of 18 participants will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women at high risk for breast cancer, defined by at least 1 of the following criteria:

  * Projected 5-year probability of invasive breast cancer at least 1.66%, as determined by the Breast Cancer Risk Assessment Tool
  * Prior node-negative breast cancer
  * Prior biopsy indicating atypical lobular or ductal hyperplasia or carcinoma in situ
  * Age 60 and over
* Non-smoker confirmed by urine cotinine test
* No concurrent breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Sex:

* Female

Menopausal status:

* Premenopausal (regular menstrual cycles of 24-36 days within the past 6 months) OR
* Postmenopausal (no menstrual cycle for at least 6 months)

Performance status:

* Not specified

Life expectancy:

* At least 1 year

Hematopoietic:

* Absolute granulocyte count greater than 1,500/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin less than 1.8 mg/dL
* Aspartate aminotransferase (AST) and Alanine transaminase (ALT) less than 110 U/L
* Alkaline phosphatase less than 300 U/L
* Albumin greater than 3 g/dL

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* No acute or unstable cardiovascular condition based on electrocardiogram

Other:

* Mild seasonal allergies allowed
* No serious or life-threatening drug allergies
* No other serious intolerances or allergies
* No more than 20% above or below ideal body weight
* No acute or unstable medical condition by physical examination or laboratory tests
* No chronic headaches, dysphoria, fatigue, dizziness, blurred vision, insomnia, rhinorrhea, nausea, vomiting, abdominal pain, diarrhea, constipation, or similar conditions
* No serious illness requiring chronic drug therapy
* No active malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception 1 month before, during, and for 1 month after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* At least 2 months since prior hormonal therapy as contraception or hormone replacement therapy (HRT)
* No concurrent sex hormones as contraception for premenopausal women
* No concurrent HRT for postmenopausal women

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 6 months since prior investigational drugs
* At least 1 month since prior weekly consumption of more than 3 medium servings (half cup each) of cruciferous vegetables
* No concurrent vegetarian diet or weekly consumption of more than 3 medium servings (half cup each) of cruciferous vegetables
* No continuous supplement intake
* No recent change in medications or dosage of medications

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-01; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aryeh Hurwitz, MD, Study Chair — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States